CLINICAL TRIAL: NCT07031882
Title: Liberty Analyzer WBC System: Reference Interval Study
Acronym: REFINE
Status: Not yet recruiting | Type: Observational
Sponsor: Entia Ltd (Industry)
Responsible Party: Sponsor
Other Study IDs: CTM-PRO-00174
Record Dates: First submitted 2025-05-29; First posted 2025-06-22 (Actual); Last update posted 2025-06-22 (Actual); Status verified 2025-06

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | Unapproved Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Healthy volunteers
  Interventions: Device: Liberty Analyzer WBC System

INTERVENTIONS:
Device: Liberty Analyzer WBC System — Participants will donate capillary samples to be analysed by the Liberty Analyzer System WBC

SUMMARY:
The purpose of this study is to establish the reference intervals for WBC and granulocytes for the Liberty Analyzer WBC System.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥21 years old at the time of study entry
* Able to provide written informed consent

Exclusion Criteria:

* Inadequate use and understanding of the English language, requiring a translator
* Undergone tattooing or body piercing within the 7 days prior to the study visit
* Undergone vaccination within the 7 days prior to the study visit
* Episode of upper respiratory infection within the 30 days prior to the study visit
* Use of oral corticosteroid medications within the 30 days prior to the study visit
* Undergone surgery within the 90 days prior to the study visit
* Been hospitalised within the 90 days prior to the study visit
* Donated blood or plasma within the 90 days prior to the study visit
* Pregnant at the time of the study visit
* Breastfeeding at the time of the study visit
* Current diagnosis of anemia (including iron deficiency anemia, vitamin deficiency anemia, aplastic anemia and/or hemolytic anemia)
* Current diagnosis of high blood pressure
* Current diagnosis of diabetes mellitus
* History or current diagnosis of chronic kidney disease or end-stage renal disease
* History or current diagnosis of cancer
* History or current diagnosis of cardiovascular disease
* History or current use of radiotherapy of the chest or abdomen
* History or current diagnosis of the following conditions known to affect the CBC differential count:
* Immune Thrombocytopenic Purpura (ITP)
* Systemic Lupus Erythematosus (SLE)
* Rheumatoid Arthritis (RA)
* Antiphospholipid Syndrome (APS)
* Sjogren's Syndrome
* Tuberculosis (TB)
* HIV
* Hepatitis B/C
* G6PD Deficiency
* Sickle Cell Disease/Trait
* Inflammatory Bowel Disease (IBD)
* Eptein Barr virus
* CMV Cytomegalovirus
* Myelodysplastic Syndromes (MDS) / CMML
* Asplenia

Participants who meet the following criteria will be excluded a posteriori:

* Hemoglobin, hematocrit, red cell and/or total white blood cell count obtained by standard laboratory analysis of the participant's venous blood sample, that fall(s) outside of the applicable reference interval(s) in use at the study site.
* Iron, ferritin, transferrin, total Iron Binding Capacity (TIBC) and/or transferrin saturation results obtained by standard laboratory analysis of the participant's venous blood sample, that fall(s) outside of the applicable reference interval(s) in use at the study site.
* Alanine aminotransferase (ALT), aspartate aminotransferase ( AST), alkaline phosphatase (ALP), gamma-glutamyl transferase (GGT), total bilirubin, conjugated bilirubin, albumin and/or total protein results obtained by standard laboratory analysis of the participant's venous blood sample, that fall(s) outside of the applicable reference interval(s) in use at the study site.
* Creatinine, estimated glomerular filtration rate (eGFR), blood urea nitrogen (BUN), sodium, potassium, chloride and/or bicarbonate results obtained by standard laboratory analysis of the participant's venous blood sample, that fall(s) outside of the applicable reference interval(s) in use at the study site.
* C-reactive protein (CRP) results obtained by standard laboratory analysis of the participant's venous blood sample, that fall outside of the applicable reference interval in use at the study site.
* Self-report to be taking medication(s) that are subsequently identified as interfering substances for the Liberty Analyzer WBC System

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Non-diseased adults.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
To establish the 95% reference interval for WBC for the Liberty Analyzer WBC System, reported with 90% confidence intervals. | Through study completion, an average of 1 day
To establish the 95% reference interval for absolute granulocytes for the Liberty Analyzer WBC System, reported with 90% confidence intervals. | Through study completion, an average of 1 day

IPD SHARING:
Plan to Share IPD: Undecided
To be determined by study management group.